CLINICAL TRIAL: NCT05479747
Title: The Effect of Trypsin-Chymotrypsin On Postoperative Pain After Single Visit Endodontic Treatment A Randomized Controlled Trial
Brief Title: Efficacy of Trypsin-Chymotrypsin On Post-operative Pain After Single Visit Root Canal Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa Adly Abd El-Sattar Mahmoud, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-Rec IM012110
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: Effect of Drug
Keywords: Trypsin and chymotrypsin; Ibuprofen; postoperative pain; Analgesic drugs; pain control drugs
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ibuprofen (Brufen) (Active Comparator): Participants were handed Brufen (Ibuprofen) (Abbott chemical laboratories, Advil, USA) 600 mg 3 times daily for 3 days after meals in tightly sealed envelope with an included written paper contained the instruction for dose administration.
  Interventions: Drug: post operative analgesics
- Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) (Experimental): Participants were handed Ambezim G (Trypsin 5 mg Chymotrypsin 5 mg) (Global Napi Pharmaceutical Company, Giza, Egypt) 3 times daily for 3 days one hour before meals in tightly sealed envelope with an included written paper contained the instruction for dose administration.
  Interventions: Drug: post operative analgesics
- Ibuprofen (Brufen) + Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) (Active Comparator): Participants were handed Brufen (Ibuprofen) (Abbott chemical laboratories, Advil, USA) 600 mg 3 times daily for 3 days after meals and Ambezim G (Trypsin 5 mg Chymotrypsin 5 mg) (Global Napi Pharmaceutical Company, Giza, Egypt) 3 times daily for 3 days one hour before meals in tightly sealed envelope with an included written paper contained the instruction for dose administration.
  Interventions: Drug: post operative analgesics
- Placebo pills (Sugar pills) (Placebo Comparator): Participants were handed postoperatively sugar pills (Placebo pills) (Department of pharmaceutics & industrial pharmacy at Faculty of pharmacy Ain Shams University, Cairo, Egypt) 3 times daily for 3 days in tightly sealed envelope with an included written paper contained the instruction for dose administration.
  Interventions: Drug: post operative analgesics

INTERVENTIONS:
Drug: post operative analgesics — post-operative pain killer
  Other Names: pain control drug

SUMMARY:
Achieving effective pain control after endodontic treatment is still a disruptive event to all the clinicians. There is a knowledge gap regarding the effect of protease on postoperative pain following root canal treatment, therefore, the efficacy of Trypsin-Chymotrypsin on post endodontic pain was evaluated clinically in a randomized triple-blind trial.

DETAILED DESCRIPTION:
This study approved by the institutional review of board (IRB) of the ethics committee at the Faculty of Dentistry, Ain Shams University, Cairo, Egypt under approval number FDASU-Rec IM012110.

This study design was a prospective, parallel triple blind phase IV randomized clinical trial.

A pilot study was performed on five patients in each group and its results were used for sample size calculation. Based upon the results of the pilot study; the minimum estimated sample size was a total of 52 patients. Sample size was increased to 60 for compensation of the drop-out. Sample size calculation was performed by using G*Power Version 3.1.9.2.

All included patient signed an informed consent prior to start of the study.

Randomization and blinding:60 patients who had the eligibility criteria were allocated randomly according to the ratio of 1:1 to each group. Randomization was performed by using computer software (www.randome.org).

Allocation concealment mechanism: Random sequence generations, allocation concealment and interventions preparation were occurred before starting by the help of one independent person who concealed the allocation sequence from the investigators in opaque and tightly sealed envelope. Before study implementation, this person also divided the medicaments into 60 tightly sealed opaque envelopes contained a treatment with the recommended dose and labeled by one-digit alphabetical symbol (X, Y, Z, R).

Implementation of the study: After root canal treatment, post-operative medicaments were assigned by telephone verification. This independent person informed the operator which drug should be prescribed in the form of X, Y, Z or R to maintain operator blinding. The investigators used the computerized generated randomization protocol for each eligible patient. So, patients were enrolled into each of the groups and prescribed with different post-operative intervention. All pain assessment forms and data were monitored by a trained clinician. He was not a part of the study team.The statistician was also blinded.

Patient history revealed diffuse lingering pulpal pain. Cold sensibility testing with Endo-Ice (1,1,1,2 Tetrafluoroethane; Hygenic Corp) indicated a moderate to severe response. Vitality was matched with the contra lateral as control. The vitality was established clinically by blood observation in the canal. Teeth had no sensitivity to percussion or palpation. Radiographically had normal periapical condition. Endodontic treatment procedures were done by the same operator in the post-graduate clinic of the Endodontic Department of the Faculty of Dentistry, Ain Shams University, Egypt. Patients were assessed by a trained clinician who was not a part of the study team.

85 patients were assessed for the eligibility criteria. 25 individuals were excluded due to different reasons. 60 participants were included. They were randomized into four groups (N = 15).

Group I: (ibuprofen) Participants were given ibuprofen 600 mg 3 times per day for 3 days after each of the three meals.

Group II: (Trypsin-Chymotrypsin) Participants were given (Trypsin 5 mg Chymotrypsin 5 mg3 times per day for 3 days one hour before each of the three meals.

Group III: (ibuprofen + Trypsin Chymotrypsin) Participants were given ibuprofen 600 mg 3 times per day for 3 days after each of the three meals and (Trypsin 5 mg Chymotrypsin 5 mg) 3 times per day for 3 days one hour before each of the three meals.

Group IV: (placebo) Participants were given postoperatively placebo sugar pills 3 times per day for 3 day.

All participant were asked to record their postoperative pain intensity at 6h ,12h ,24h, 48h ,72h following obturation. They also asked to report the occurrence of any side effects.

Data analysis:

Statistical analysis was undertaken with IBM SPSS Statistics. Age difference was analyzed by using one-way ANOVA test. For Pain records, Kruskal-Wallis test for comparison among the four groups, Friedman's test for changes by time intervals in each group and for pair-wise comparisons when Kruskal-Wallis or Friedman's test was significant, Dunn's test was used. Chi-square test was used for qualitative data. The significance level was set at P ≤ 0.05.

ELIGIBILITY:
Inclusion criteria:

* Egyptian healthy symptomatic both gender patients
* aged (18- 40) years old
* with no physical disability, facial paresthesia or psychological problems
* had mandibular first molars with symptomatic irreversible pulpitis and with normal appearance radiographically.

Exclusion criteria:

* The vulnerable group
* participants who un abled to read and fill the questionnaire,
* those who took preoperative analgesics 24 h prior to treatment
* those with known sensitivity to the drugs used in this study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Hashem, PHD, Study Chair — Head of endodontic department Faculty of dentistry Ain Shams University, cairo,Egypt; Tariq Y Abdel Rahman, PHD, Study Director — Lecturer, Endodontic Department, Faculty of Dentistry, Ain Shams University; Alaa A Abd El Sattar, Master, Principal Investigator — Faculty of Dentistry, Ain Shams University
Locations (1):
- Ahmed Abdel Rahman Hashem, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hashem AAR, Abd El Sattar AA, Abdel Rahman TY. The Effect of Trypsin-Chymotrypsin on Postoperative Pain after Single Visit Endodontic Treatment: A Randomized Controlled Trial. J Endod. 2023 Mar;49(3):240-247. doi: 10.1016/j.joen.2022.12.010. Epub 2022 Dec 24. PMID 36574828

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibuprofen (Brufen) | Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Ibuprofen (Brufen) + Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Placebo Pills (Sugar Pills)
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen (Brufen) | Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Ibuprofen (Brufen) + Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Placebo Pills (Sugar Pills) | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (8) | 27.8 (8) | 27.9 (8.1) | 28 (7.7) | 27.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 9 | 8 | 32
  Male | 7 | 8 | 6 | 7 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Egyptian | 15 | 15 | 15 | 15 | 60
Region of Enrollment [Number; unit: participants]
  Egypt | 15 | 15 | 15 | 15 | 60
pre-operative pain scores [Mean (Standard Deviation); unit: units on a scale] — Pre-operative pain scores was assessed by using a Numeric Rating Scale (NRS). The minimum score value is zero. The maximum score value is ten. Maximum scores indicate the worst possible outcome.
  units on a scale | 8.4 (0.63) | 8.53 (1.13) | 8.13 (1.36) | 8.73 (0.8) | 8.4 (0.98)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Trypsin-Chymotrypsin on Post-operative Pain After Single Endodontic Treatment in Teeth With Symptomatic Irreversible Pulpitis
Description: analgesic effect assessed by numerical rating scale. The minimum score value is zero. The maximum score value is ten. Maximum scores indicate the worst possible outcome.
Time Frame: from 6 hours following drug intake after obturation to 72 hours (start with 6 hours first interval then at 12 hours intervals)
Population: We detect the effect of Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) on post-operative pain and compared its effect with the most known potent analgesic ibuprofen (Brufen) and with a combination of both drugs and with Placebo pills (Sugar pills) for better evaluation of its efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen (Brufen) | Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Ibuprofen (Brufen) + Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Placebo Pills (Sugar Pills)
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale
  after 6 hours follow up | 3.47 (1.55) | 3.53 (1.46) | 2.93 (1.33) | 6.13 (0.64)
  after 12 hours follow up | 2 (1.41) | 1.87 (1.51) | 1.4 (0.91) | 4.47 (0.64)
  after 24 hours follow up | 0.87 (1.06) | 0.8 (1.08) | 0.2 (0.41) | 3.4 (0.74)
  after 48 hours follow up | 0 (0) | 0.13 (0.52) | 0 (0) | 2.47 (0.64)
  after 72 hours follow up | 0 (0) | 0.13 (0.52) | 0 (0) | 1.2 (0.77)

2. Secondary Outcome: Synergistic Effect With NSAIDS
Description: as for outcome 1
Time Frame: as for outcome 1
Population: We compared the result of each pharmaceutical alone with the result of a combination of both drugs in group Ibuprofen (Brufen) + Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) to conclude the secondary outcome (synergistic effect with NSAIDS).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen (Brufen) | Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Ibuprofen (Brufen) + Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Placebo Pills (Sugar Pills)
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale
  after 6 hours follow up | 3.47 (1.55) | 3.53 (1.46) | 2.93 (1.33) | 6.13 (0.64)
  after 12 hours follow up | 2 (1.41) | 1.87 (1.51) | 1.4 (0.91) | 4.47 (0.64)
  after 24 hours follow up | 0.87 (1.06) | 0.8 (1.08) | 0.2 (0.41) | 3.4 (0.74)
  after 48 hours follow up | 0 (0) | 0.13 (0.52) | 0 (0) | 2.47 (0.64)
  after 72 hours follow up | 0 (0) | 0.13 (0.52) | 0 (0) | 1.2 (0.77)

3. Secondary Outcome: Reported Side Effect
Description: assessed by Passive surveillance of harm. It depends on adverse effects reported by the participants.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: reported side effects
Arm/Group | Ibuprofen (Brufen) | Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Ibuprofen (Brufen) + Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Placebo Pills (Sugar Pills)
Number analyzed (Participants) | 15 | 15 | 15 | 15
reported side effects
  after 6 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  after 12 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  after 24 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  after 48 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  after 72 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: from 6 hours following drug intake after obturation to 72 hours (start with 6 hours first interval then at 12 hours intervals)
Description: Only healthy individuals and those with no sensitivity to pharmaceuticals used in our study participated in the trial, so they were not liable for any adverse effects.
  Even no one complained about the possible side effects of these pharmaceuticals.
Arm/Group | Ibuprofen (Brufen) | Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Ibuprofen (Brufen) + Trypsin 5 mg Chymotrypsin 5 mg (Ambezim G) | Placebo Pills (Sugar Pills)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT05479747/Prot_SAP_000.pdf